CLINICAL TRIAL: NCT01320033
Title: A Multi Center, Randomized, Double Blind, Placebo Controlled, 3 Arm, Parallel Group Study Comparing the Efficacy and Safety of CD2475/101 40 mg Tablets Versus Placebo and Doxycycline 100 mg Capsules Once Daily in the Treatment of Inflammatory Lesions in Subjects With Acne Vulgaris
Brief Title: Placebo Controlled Efficacy and Safety Study of CD2475/101 40 mg Tablets vs. Placebo and Doxycycline 100 mg Capsules Once Daily in the Treatment of Inflammatory Lesions of Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18195
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2019-12

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; inflammatory lesions
MeSH Terms: conditions — Acne Vulgaris | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CD2475/101 40 mg (Experimental): Participants receive 40 mg of CD2475/101 oral tablet plus placebo capsule orally once daily for 16 weeks.
  Interventions: Drug: CD2475/101 40 mg; Drug: Placebo
- Doxycycline 100 mg (Active Comparator): Participants receive 100 mg of Doxycycline capsule plus placebo tablet orally once daily for 16 weeks.
  Interventions: Drug: Doxycycline 100 mg; Drug: Placebo
- Placebo (Placebo Comparator): Participants receive matching placebo tablet plus placebo capsule orally once daily for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CD2475/101 40 mg — Participants receive 40 mg of CD2475/101 tablets once a day for 16 weeks.
  Arms: CD2475/101 40 mg
Drug: Doxycycline 100 mg — Participants receive 100 mg of Doxycycline capsule once a day for 16 weeks
  Arms: Doxycycline 100 mg
Drug: Placebo — Participants receive matching placebo tablet, matching placebo capsule once a day for 16 weeks.

SUMMARY:
The primary objectives of the study is to show CD2475/101 40mg tablets taken once a day for 16 weeks is superior to the placebo in Change from baseline to Week 16(Last Observation Carry Forward, Intent To Treat) in inflammatory lesion counts.

DETAILED DESCRIPTION:
Investigator's global assessment and lesion count will be performed at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 12 years of age or older
* acne vulgaris with facial involvement
* A score of 3 (Moderate) or 4 (Severe) on the Investigator's Global Assessment Scale (inflammatory)
* 25 to 75 inflammatory lesions (papules and pustules) on the face (including the nose)

Exclusion Criteria:

* More than two acne nodules/cysts on the face
* Acne conglobata, acne fulminans, secondary acne (chloracne, drug induced acne, etc.), or severe acne requiring systemic retinoid treatment
* Underlying diseases or other dermatologic conditions that require the use of interfering topical or systemic therapy such as, but not limited to, atopic dermatitis, perioral dermatitis or rosacea
* Beard or facial hair which might interfere with study assessments
* planning excessive exposure to sun or ultraviolet light during the study (i.e. natural or artificial sunlight, including tanning booths and sun lamp)
* Use of oral contraceptives solely for control of acne
* Liver function test alanine transaminase (ALT) and/or aspartate transaminase (AST) 2.5 times above upper limit of normal
* Renal function test serum creatinine at 150 umol/L (17 mg/L) or higher
* Presence of oral or genital candidiasis or history of multiple episodes of oral or genital candidiasis
* Females who intend to conceive a child within 5 months following Baseline visit
* Males who intend to conceive a child with partner during the study period
* Requiring concomitant use of methoxyflurane

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2011-03-29 (Actual); Primary Completion 2012-01-03 (Actual); Study Completion 2012-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D
Locations (31):
- United States (31):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Dermatology Research Associates, Inc., Los Angeles, California
  - Colorado Medical Research Center, Denver, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - International Dermatology Research, Inc., Miami, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Dermatology Specialists PC, Louisville, Kentucky
  - Somerset Skin Care Center, Troy, Michigan
  - Grekin Skin Care, Warren, Michigan
  - Central Dermatology, PC, St Louis, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - Academic Dermatology, Albuquerque, New Mexico
  - Helendale Dermatology & Medical Spa, Rochester, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Haber Dermatology & cosmetic Surgery, Inc, South Euclid, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Oregon Dermatology & Research Center, Portland, Oregon
  - Stephen Schleicher, Hazleton, Pennsylvania
  - Palmetto Clinical Trial Services, LLC, Greenville, South Carolina
  - Dermatology Research Associates, Nashville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - Derm Research, Inc, Austin, Texas
  - J&S Studies, College Station, Texas
  - Suzanne Bruce and associates P.A. The Center for skin Research, Houston, Texas
  - Center for Clinical Studies, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Stephen Miller MD, San Antonio, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - Premier Clinical Research, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in United States between 29 March 2011 (first participant first visit) to 3 January 2012 (last participant last visit).
Pre-assignment Details: A total of 662 participants randomized the study and dispensed with study drug out of which 487 completed study.
Groups:
- CD2475/101 40 mg: Participants received 40 milligrams (mg) of CD2475/101 oral tablet plus placebo capsule orally once daily for 16 weeks.
- Doxycycline 100 mg: Participants received 100 mg of Doxycycline capsule plus placebo tablet orally once daily for 16 weeks.
- Placebo: Participants received matching placebo tablet plus placebo capsule orally once daily for 16 weeks.
Period: Overall Study
Arm/Group | CD2475/101 40 mg | Doxycycline 100 mg | Placebo
Started | 216 | 224 | 222
Completed | 158 | 160 | 169
Not Completed | 58 | 64 | 53
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Adverse Event | 9 | 7 | 8
Not completed — Withdrawal by Subject | 22 | 23 | 23
Not completed — Protocol Violation | 3 | 5 | 3
Not completed — Lost to Follow-up | 22 | 26 | 17
Not completed — Other | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population consisted of all participants who were randomized and to whom study drug was dispensed.
Groups:
- CD2475/101 40 mg: Participants received 40 mg of CD2475/101 oral tablet plus placebo capsule orally once daily for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | CD2475/101 40 mg | Doxycycline 100 mg | Placebo | Total
Number analyzed (Participants) | 216 | 224 | 222 | 662
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 123 | 132 | 133 | 388
  Between 18 and 65 years | 93 | 92 | 89 | 274
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.6 (7.70) | 19.6 (7.54) | 18.7 (6.34) | 19.3 (7.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 121 | 115 | 351
  Male | 101 | 103 | 107 | 311
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 30 | 37 | 102
  Not Hispanic or Latino | 181 | 194 | 185 | 560
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 7 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 47 | 49 | 40 | 136
  White | 159 | 163 | 170 | 492
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 216 | 224 | 222 | 662

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Inflammatory Lesion Counts to Week 16 (Last Observation Carried Forward [LOCF])
Description: The Inflammatory lesion count was the count of papules and pustules: papule was a small, solid elevation less than 0.5 cm in diameter, pustule was a small, circumscribed elevation of the skin that contains yellow-white exudate. Change from baseline in inflammatory lesion counts to Week 16 (LOCF) were reported.
Time Frame: From Baseline up to Week 16 (LOCF)
Population: Intent To Treat (ITT) population consisted of all participants who were randomized and to whom study drug was dispensed.
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | CD2475/101 40 mg | Doxycycline 100 mg | Placebo
Number analyzed (Participants) | 216 | 224 | 222
lesion count | -16.1 (11.39) | -12.9 (14.60) | -12.6 (16.44)
Statistical Analysis 1: Comparison: CD2475/101 40 mg vs Placebo; Test type: Superiority; p = 0.006, ANCOVA; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-6.1 to -1.1]
Statistical Analysis 2: Comparison: CD2475/101 40 mg vs Doxycycline 100 mg; Test type: Superiority; p = 0.024, ANCOVA; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-5.4 to -0.4]
Statistical Analysis 3: Comparison: Doxycycline 100 mg vs Placebo; Test type: Superiority; p = 0.595, ANCOVA; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-3.2 to 1.8]

2. Secondary Outcome: Investigator Global Assessment (IGA) Success Rate at Week 16 (Last Observation Carried Forward [LOCF])
Description: IGA scale consisted of 5 grades (0-4) among which 0= Clear (no evidence of papules or pustules [inflammatory lesions]), 1= Almost clear (rare non-inflamed papules (papules must be resolving and hyperpigmented, though not pink-red), 2= Mild (few inflammatory lesions [papules/pustules only; no nodulo-cystic lesions]), 3=Moderate (multiple inflammatory lesions evident: many papules/pustules; up to two nodulocystic lesions), 4= Severe (inflammatory lesions are more apparent, many papules/pustules, few nodulo-cystic lesions). Success rate was defined as percentage of participants who achieved an Investigator Global Assessment (IGA) score of 1 (almost clear) or 0 (Clear) and at least a 2-grade improvement from Baseline to Week 16 (LOCF).
Time Frame: Week 16 (LOCF)
Population: ITT Population consisted of all participants who were randomized and to whom study drug was dispensed.
Measure: Number; unit: Percentage of participants
Arm/Group | CD2475/101 40 mg | Doxycycline 100 mg | Placebo
Number analyzed (Participants) | 216 | 224 | 222
Percentage of participants | 14.4 | 13.8 | 7.7

3. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Counts to Week 16 (Last Observation Carried Forward [LOCF])
Description: The Inflammatory lesion count was the count of papules and pustules: papule was a small, solid elevation less than 0.5 cm in diameter, pustule was a small, circumscribed elevation of the skin that contains yellow-white exudate. Percent change from baseline in inflammatory lesion counts to Week 16 (LOCF) were reported.
Time Frame: From Baseline up to Week 16 (LOCF)
Population: ITT population consisted of all participants who were randomized and to whom study drug was dispensed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CD2475/101 40 mg | Doxycycline 100 mg | Placebo
Number analyzed (Participants) | 216 | 224 | 222
percent change | -48.6 (31.72) | -40.3 (40.90) | -37.1 (44.45)

4. Secondary Outcome: Percent Change From Baseline in Total Lesion Counts to Week 16 (Last Observation Carried Forward [LOCF])
Description: Total lesions were the sum of inflammatory lesion counts, non-inflammatory lesion counts, nodules and cysts. Percentage change from baseline in total lesion counts to Week 16 were reported.
Time Frame: From Baseline up to Week 16 (LOCF)
Population: ITT population consisted of all participants who were randomized and to whom study drug was dispensed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CD2475/101 40 mg | Doxycycline 100 mg | Placebo
Number analyzed (Participants) | 216 | 224 | 222
percent change | -38.3 (32.24) | -27.8 (43.94) | -27.8 (38.05)

5. Secondary Outcome: Change From Baseline in Non-Inflammatory Lesion Counts to Week 16 (Last Observation Carried Forward [LOCF])
Description: The non-inflammatory lesion count was the count of open and closed comedones: Open comedone was a pigmented dilated pilosebaceous orifice (blackhead). Closed comedone was a tiny white papule (whitehead). Change from baseline in non-inflammatory lesion counts to week 16 were reported
Time Frame: From Baseline up to Week 16 (LOCF)
Population: ITT population consisted of all participants who were randomized and to whom study drug was dispensed.
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | CD2475/101 40 mg | Doxycycline 100 mg | Placebo
Number analyzed (Participants) | 216 | 224 | 222
lesion count | -10.0 (21.49) | -5.2 (21.60) | -5.8 (18.19)

6. Secondary Outcome: Global Assessment for Inflammatory Lesions of Truncal Acne at Baseline, Week 12, and Week 16
Description: Global assessments for inflammatory lesions of truncal acne were done separately on back and chest. The global assessments severity scale included 5 grades (0-4): where in 0= Clear-no evidence of papules or pustules (inflammatory lesions), 1= Almost clear- rare non-inflamed papules (papules must be resolving and may be hyperpigmented, though not pink-red), 2=Mild- few inflammatory lesions (papules/pustules only; no nodulo-cystic lesions), 3=Moderate- multiple inflammatory lesions evident: many papules/pustules; may be a few nodulocystic lesions, 4=Severe- inflammatory lesions are more apparent, many papules/pustules, may be a few nodulo-cystic lesions.
Time Frame: Baseline, Week 12, and Week 16
Population: ITT population consisted of all participants who were randomized and to whom study drug was dispensed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CD2475/101 40 mg | Doxycycline 100 mg | Placebo
Number analyzed (Participants) | 216 | 224 | 222
Units on a scale
  Baseline : Lesion of Truncal Acne on Back | 1.6 (1.10) | 1.5 (1.09) | 1.5 (1.07)
  Baseline : Lesion of Truncal Acne on Chest | 1.2 (1.04) | 1.2 (1.00) | 1.1 (0.98)
  Week 12 : Lesions of Truncal Acne on Back | 1.2 (1.06) | 1.1 (1.05) | 1.2 (1.04)
  Week 12 : Lesion of Truncal Acne on Chest | 0.9 (0.94) | 0.9 (0.99) | 0.9 (0.95)
  Week 16 : Lesions of Truncal Acne on Back | 1.1 (1.06) | 1.0 (1.06) | 1.2 (1.03)
  Week 16 : Lesion of Truncal Acne on Chest | 0.9 (1.01) | 0.8 (0.93) | 0.9 (0.95)

7. Secondary Outcome: Number of Participants With at Least One Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participants administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Number of participants with at least one AE were reported.
Time Frame: From Baseline up to Week 16
Population: Safety Population consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CD2475/101 40 mg | Doxycycline 100 mg | Placebo
Number analyzed (Participants) | 216 | 223 | 222
Participants | 63 | 83 | 89

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 16
Groups:
- Placebo: Participants received 100 mg of Doxycycline capsule plus placebo tablet orally once daily for 16 weeks.
Arm/Group | CD2475/101 40 mg | Doxycycline 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/216 | 0/223 | 0/222
Serious Adverse Events (participants affected / at risk) | 1/216 | 4/223 | 2/222
Other Adverse Events (participants affected / at risk) | 29/216 | 51/223 | 29/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD2475/101 40 mg (N=216) | Doxycycline 100 mg (N=223) | Placebo (N=222)
Affective disorder (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple drug overdose intentional (Injury, poisoning and procedural complications) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CD2475/101 40 mg (N=216) | Doxycycline 100 mg (N=223) | Placebo (N=222)
Nasopharyngitis (Infections and infestations) | 7 | 7 | 14
Headache (Nervous system disorders) | 14 | 15 | 6
Nausea (Gastrointestinal disorders) | 7 | 14 | 4
Vomiting (Gastrointestinal disorders) | 1 | 15 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes